CLINICAL TRIAL: NCT02978872
Title: Comparison of Coagulation Parameters in Arterial and Venous Blood Measured Using the Quantra System
Brief Title: Quantra Determination of Coagulation Parameters in Arterial and Venous Blood
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: HEMCS-005
Record Dates: First submitted 2016-11-28; First posted 2016-12-01 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Surgery
Keywords: Cardiac surgery; Quantra; Viscoelastic testing; Coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Quantra™ System is a novel point-of-care diagnostic device designed to perform whole blood coagulation analysis. This study compares Quantra measurements determined in arterial versus venous blood samples obtained from patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which utilizes SEER Sonorheometry, an ultrasound-based technology, to characterize the dynamic changes in the viscoelastic properties of a blood sample during coagulation and clot lysis. Viscoelastic testing performed using existing technologies is typically performed on arterial samples obtained from patients undergoing surgical procedures, although reference ranges for these tests have been established for venous blood only.

The aim of this study is to evaluate potential differences between Quantra measurements determined in arterial versus venous blood samples obtained from patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for cardiac surgery, utilizing cardiopulmonary bypass, or including placement of a ventricular assist device
* Subject is ≥18 years
* Subject is willing to participate and he/she has signed a consent form
* Subject may participate if they have a history of bleeding or are on preoperative anticoagulant therapy

Exclusion Criteria:

* Subject is unable to provide written informed consent
* Subject is younger than 18 years
* Subject is incarcerated at the time of the study
* Subject is currently enrolled in a study that may confound the results of the proposed study
* Subject is affected by a condition that, in the opinion of the surgical team, may pose additional risks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for cardiac surgery, utilizing cardiopulmonary bypass, or including placement of a ventricular assist device.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Clot Time and Clot Stiffness results between arterial and venous samples | Up to 24 hours
  Coagulation function assessed by Quantra at 2 time points (Baseline and either during cardiac bypass or post-bypass)

SECONDARY OUTCOMES:
Comparison of Quantra results to standard coagulation test results in venous samples | Up to 24 hours
  Coagulation function assessed by Quantra and standard coagulation tests at 2 time points (Baseline and either during cardiac bypass or post-bypass)
Comparison of Quantra results to comparable ROTEM results in venous samples | Up to 24 hours
  Coagulation function assessed by Quantra and ROTEM at 2 time points (Baseline and either during cardiac bypass or post-bypass)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No